CLINICAL TRIAL: NCT03068871
Title: A Comparison of Two Psycho-educational Group Interventions for Tinnitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0841-16-TLV
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CET (Experimental): CET - Coping Effectiveness Training group.
  Interventions: Other: CET
- ACT (Experimental): ACT - Acceptance and Commitment Therapy group
  Interventions: Other: ACT

INTERVENTIONS:
Other: ACT — Psycho-educational group
  Arms: ACT
Other: CET — Psycho-educational group
  Arms: CET

SUMMARY:
participants will be randomized into one of three groups: 3-session CET intervention, 3-session ACT intervention, or Waiting List group. Each weekly session will last up to 2 hours and 10 participants will be assigned to each group. There will be two cohorts, with 30 participants in each cohort. The Waiting List group will receive the CET intervention after the groups have completed theirs.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus lasting more than 3 months
* Hebrew speaking
* Use hearing aids if needed
* Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
COPE | Before the intervention (T1) and at the end of intervention (T2-4 weeks after T1), 1 month after end of intervention (T3)
  Coping scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Centre, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided